CLINICAL TRIAL: NCT02482272
Title: Efficacy and Safety of Continuing Lamivudine Plus Adefovir or Adefovir Versus Switching to Entecavir Plus Adefovir in Patients With Chronic Hepatitis B Who Have Resistant Mutants to Lamivudine and Show Suboptimal Response to Combination of Lamivudine Plus Adefovir or Adefovir Monotherapy
Brief Title: Compare Continuing Lamivudine Plus Adefovir or Adefovir Versus Switching to Entecavir Plus Adefovir in Patients With LAM-resistant Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Hwa Chung, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENTADE
Record Dates: First submitted 2015-06-01; First posted 2015-06-26 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; adefovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamivudine plus Adefovir or Adefovir (Active Comparator): Lamivudine+Adefovir or Adefovir for 48 weeks
  Interventions: Drug: Lamivudine; Drug: Adefovir
- Entecavir plus Adefovir (Experimental): Entecavir+Adefovir for 48 weeks
  Interventions: Drug: Adefovir; Drug: Entecavir

INTERVENTIONS:
Drug: Lamivudine — Lamivudine 100mg/day orally
  Arms: Lamivudine plus Adefovir or Adefovir
Drug: Adefovir — Adefovir 10mg/day orally
Drug: Entecavir — Entecavir 1mg/day orally
  Arms: Entecavir plus Adefovir

SUMMARY:
The purpose of this study is to compare efficacy and safety of continuing Lamivudine plus Adefovir or Adefovir versus switching to Entecavir plus Adefovir in patients with LAM-resistant chronic hepatitis B who have suboptimal response to Lamivudine plus Adefovir or Adefovir

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B
* Age ≥ 20 year old
* Currently taking Lamivudine and Adefovir combination therapy or Adefovir monotherapy for chronic HBV infection for 24 weeks
* Proven Lamivudine resistant mutation
* HBV DNA levels at screening ≥ 15 IU/mL
* Females must be post-menopausal, unable to conceive, or test negative for pregnancy via urine test
* Patient is able to give written informed consent prior to study start and to comply with the study requirements

Exclusion Criteria:

* A history or current of decompensated cirrhosis or hepatocellular carcinoma
* Currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy
* Co-infected with HCV or HIV
* A history of organ transplantation
* Pregnant or breast-feeding
* Current clinically relevant of abuse of alcohol or drugs.
* Significant immunocompromised, gastrointestinal, renal(serum creatinine ≥ 1.5 mg/dL), hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic, allergic disease or medical illness that in the investigator's opinion might interfere with therapy
* malignancy in previous 5 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA<15IU/mL | week 48

SECONDARY OUTCOMES:
Proportion of patients with HBV DNA<15IU/mL | Day1, week12, week 24, week 36, week 48
The change of HBV DNA from the baseline | week 48
Proportion of patients with ALT normalization | Day1, week12, week 24, week 36, week 48
Proportion of patients with HBeAg loss and/or seroconversion | Day1, week12, week 24, week 36, week 48
The change of HBsAg from the baseline | week 48
Proportion of patients with HBsAg loss and/or seroconversion | week 24, week 48
Proportion of patients who experienced virologic breakthrough | week 48
Assessment the safety in all patients (composite measure of AE, labs, phys. exam, vital signs) | week 48
  Composite outcome measure consisting of multiple measures, including:
  1. Number of patients with Adverse events( including SAEs)
  2. Frequency and severity of Abnormalities in laboratory examinations; BUN, Albumin, AST, ALT,GGT, Creatinine, Hemoglobin, Hematocrit, Platelet Count, Prothrombin time
  3. Number of patients with Abnormalities in physical examinations; Eyes/Ears/Nose/Throat, Respiratory, Cardiovascular, Dermatological, Abdominal, Musculoskeletal, Other
  4. Number of patients with Abnormalities in vital signs ; pulse rate( beats per minute), Blood pressure(mmHg), Height(cm), weight(kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea